CLINICAL TRIAL: NCT05847504
Title: Successive Cohort Design to Iteratively Develop mSTARS
Brief Title: mHealth-supported Skills Training for Alcohol-Related Suicidality
Acronym: mSTARS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00113104
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Drinking; Suicide
MeSH Terms: conditions — Alcohol Drinking; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mSTARS (Experimental): mHealth-supported Skills Training for Alcohol-Related Suicidality, or mSTARS, is an intervention that combines a cognitive-behavioral skills training intervention in emotion regulation skills with a post-discharge mobile health (mHealth) app that encourages application of these skills to real life.
  Interventions: Behavioral: mSTARS

INTERVENTIONS:
Behavioral: mSTARS — mSTARS combines inpatient cognitive-behavioral skills training and outpatient use of a mobile app encouraging application of acquired skills to real life situations.

SUMMARY:
Suicide is a high priority public health problem and an increasingly prevalent alcohol-related consequence. One-third of people who die by suicide consume alcohol at hazardous rates in the year preceding death. Most people in an acute suicide crisis who present for treatment are admitted to acute psychiatric hospitalization. Yet, the 30-day period following discharge from hospitalization is by far the riskiest period for another suicide crisis. The specific aim for this project is to use a successive cohort design to iteratively develop an intervention called mHealth-supported Skills Training for Alcohol-Related Suicidality (mSTARS). The study team will adapt and iteratively refine a cognitive-behavioral skills training intervention in emotion regulation to be administered in an acute care setting and paired with a post-discharge mHealth app that encourages application of these skills to real life. Two cohorts of five participants each will be enrolled in the project. Participants will complete mSTARS, an intervention that combines inpatient skills training and the mHealth telephone app. Upon completion of the 30-day period, participants will complete self-report measures and participate in an interview designed to evaluate their experience with the mSTARS intervention.

DETAILED DESCRIPTION:
Suicide is a high priority public health problem and an increasingly prevalent alcohol-related consequence. One-third of people who die by suicide consume alcohol at hazardous rates in the year preceding death. Most people in an acute suicide crisis who present for treatment are admitted to acute psychiatric hospitalization. Yet, the 30-day period following discharge from hospitalization is by far the riskiest period for another suicide crisis, (post-discharge rates of suicide are 600 times the global rate). Critically, 50% of suicidal inpatients report alcohol misuse, which further heightens post-discharge risk for suicide.

Acute psychiatric hospitalization focuses on rapid crisis resolution before discharging patients back into their environments with a referral for outpatient care. Outpatient-based cognitive-behavioral skills training in emotion regulation successfully treats concurrent alcohol misuse and suicidal behavior by targeting deficits in emotion regulation associated with both behaviors. Yet, fewer than 50% of psychiatric inpatients follow up with outpatient care once discharged, and those who seek care are often unable to receive it for weeks. Persistently low use of outpatient therapies coupled with alarming post-discharge rates of suicide represents an urgent quality gap. Alternative strategies for inpatient care that extend treatment into the critical post-discharge period are clearly needed to prevent suicide in psychiatric inpatients who misuse alcohol.

The specific aim for this project is to use a successive cohort design to iteratively develop an intervention called mHealth-supported Skills Training for Alcohol-Related Suicidality (mSTARS). The study team will adapt and iteratively refine a cognitive-behavioral skills training intervention in emotion regulation to be administered in an acute care setting and paired with a post-discharge mHealth app that encourages application of these skills to real life.

Two cohorts of five participants each will be enrolled in the project. Participants will complete mSTARS, an intervention that combines inpatient skills training and the mHealth telephone app. Inpatient skills training will be completed while participants are receiving inpatient psychiatric treatment. Skills training includes content designed to improve emotional regulation skills, including motivational enhancement, emotional awareness and acceptance, thinking flexibly, changing emotions, countering cravings, and relapse prevention. Upon discharge from Duke's inpatient program, patients will download the mHealth app on their personal phones to use in the personal environments for 30 days. The app is designed to encourage participants to apply skills acquired in inpatient skills training to real-life situations. Upon completion of the 30-day period, participants will complete self-report measures and participate in a semi-structured qualitative interview designed to evaluate their experience with the mSTARS intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. hospitalized for suicide crisis at Duke BHIP
3. an AUDIT-C score indicating hazardous past-month drinking (4 for men; 3 for women) + a 90-day calendar timeline follow-back (TLFB) indicating a minimum of 3 heavy drinking days per week on average (per NIAAA standards)
4. owns a smart phone
5. fluent in English.

Exclusion Criteria:

1. current psychotic or mania symptoms indicated by the MINI Neuropsychiatric Interview 6.0.(MINI)
2. receiving ECT at the time of hospitalization, which could inhibit learning
3. engaged in weekly outpatient psychotherapy
4. discharging to another high level of psychiatric care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2028-02-04 (Estimated); Study Completion 2028-02-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants who rate the intervention a 16 or more on the Client Satisfaction Questionnaire. | 30 days
  Acceptability of treatment will be measured by an 8-item measure designed to evaluate client satisfaction. Scores range from 8 to 32, with higher scores indicating higher satisfaction.
Number of participants who score above threshold (34 or more) on the mHealth Satisfaction Questionnaire | 30 days
  Acceptability of treatment will be measured by a 14-item measure designed to measure usability of mobile health apps. Scores range from 14 to 70. Higher scores indicate higher satisfaction.
Number of participants who score 54 or more on a measure of emotion regulation skills use. | 30 days
  The Emotion Regulation Skills Questionnaire is a 27-item measure of the extent to which an individual was able to successfully use emotion regulation skills typically taught in emotion regulation skills training interventions. Scores range from 0 to 108, and higher scores indicate more successful use of emotional regulation skills.

SECONDARY OUTCOMES:
Number of participants who score above clinical range on an emotion regulation scale | 30 Days
  Emotion regulation will be measured with the Difficulties in Emotion Regulation Scale, a 36-item scale designed to evaluate emotion regulation. Scores range from 36 to 180, with higher scores indicating poorer emotion regulation. A cut score of 80 will be used.
Number of participants who score above the clinical range (T score of 70+) on the global severity index of the Symptom Checklist-90 | 30 days
  Participants will complete the Symptom Checklist-90, a self-report, 90-item measure of psychological distress with a T-score range of 30 to 120. Higher scores indicate higher distress.
Average score on the Beck Scale for Suicidal Ideation | 30 days
  Participants will complete the Beck Scale for Suicidal Ideation, a 19-item scale to assess ideation, plans, and/or intent to suicide. Scores range from 0 to 48, with higher scores indicating higher suicide risk.
Number of participants who score 40 or less on a measure of perceived efficacy to abstain from alcohol | 30 days
  Participants will complete the 20-item Alcohol Abstinence Self-Efficacy scale indicating how confident they are in ability to abstain from alcohol in certain situations. Scores range from 20 to 100, with higher scores indicating higher confidence to abstain from alcohol use.
Number of participants who score 21 or less on the Brief Inventory of Psychosocial Functioning | 30 days
  Participants will complete the 7-item Brief Inventory of Psychosocial Functioning which is a measure of how individuals are doing in their various domains of psychosocial functioning. Scores range from 0 to 49, with higher scores indicating poorer psychosocial functioning.
Average number of drinking days | 30 days
  Patients will self-report the number of drinking days in the past 30 days.
Number of participants who report re-hospitalization to an inpatient psychiatry unit. | 30 days
  Treatment inefficacy will be measured by the number of participants who are re-hospitalized in the 30 day period following their enrollment in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No